CLINICAL TRIAL: NCT01983982
Title: Effect of Chemotherapy on Pain Sensitivity and Patient-reported Symptoms in Early Stage Breast Cancer
Brief Title: Effect of Chemotherapy on Pain Sensitivity and Patient-reported Symptoms
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: Damon Runyon Cancer Research Foundation (Other)
Responsible Party: Principal Investigator, N. Lynn Henry, Assistant Professor of Internal Medicine, Medical School, University of Michigan
Other Study IDs: HUM00077174; UMCC 2013.073 (Other: University of Michigan Cancer Center)
Record Dates: First submitted 2013-11-07; First posted 2013-11-14 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Breast Cancer; Chronic Pain
Keywords: Breast Cancer; Chemotherapy; Chronic Pain; Survivorship
MeSH Terms: conditions — Breast Neoplasms; Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Adjuvant chemotherapy: Subjects will undergo pain testing, then receive standard of care chemotherapy, and then undergo pain testing.

SUMMARY:
Many breast cancer survivors report chronic pain that develops or worsens following chemotherapy. The impact of chemotherapy on the development of chronic pain is uncertain. In this proposal, we are studying the impact of chemotherapy on a patient's sensitivity to pain. We are also investigating whether a patient's sensitivity to pain is related to how many symptoms she experiences during treatment.

ELIGIBILITY:
Inclusion Criteria:

* Female gender
* Histologically proven stage I-III invasive carcinoma of the breast who is planning to receive a standard dose of adjuvant chemotherapy.
* Surgical resection should be complete at the time of study enrollment.
* Eastern Cooperative Oncology Group performance status 0-2.

Exclusion Criteria:

* Average pain over the past 24 hours of 4 or greater on a 0-10 scale.
* Peripheral sensory neuropathy grade 2 or higher.
* Personal history of schizophrenia or major depressive disorder, or history of suicidal ideation or attempt within the past 2 years.
* Thumbnail abnormalities on either hand (such as artificial nails) that are likely to alter pain perception during testing.
* Pregnant or nursing.
* No prior chemotherapy for any reason

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women initiating adjuvant chemotherapy to treat stage I-III breast cancer.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2013-11; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Feasibility of recruiting patients at chemotherapy initiation | 15 weeks
  Feasibility will be measured by the proportion of women who complete the post-chemotherapy assessment among those consenting to participate in the trial.

SECONDARY OUTCOMES:
Change in Pain Sensitivity in Breast Cancer Patients Associated with Chemotherapy | 15 weeks
  Patients will undergo quantitative sensory testing to identify change in pain threshold and in the magnitude of conditioned pain modulation before chemotherapy and shortly after the final dose of chemotherapy.
Association Between Baseline Pain-Pressure Threshold and Development of Chemotherapy-associated Acute Pain | 15 weeks
  Exploratory analyses will be conducted to examine associations between either baseline or change in quantitative sensory testing measures and change in patient-reported outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Norah L Henry, MD, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Health System, Ann Arbor, Michigan, United States